CLINICAL TRIAL: NCT01190852
Title: Single Dose Pharmacokinetics of Intranasal Azelastine Delivered by a Fixed Combination With Fluticasone in Comparison to Azelastine Nasal Sprays Single-centre, Randomised, Open-label, Three-period, Six-sequence Cross-over Trial (William's Design)
Brief Title: Single Dose Pharmacokinetics of Intranasal Azelastine Delivered by a Fixed Combination With Fluticasone in Comparison to Azelastine Nasal Sprays
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: ClinResearch, GmbH (Other); Prolytic GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: X-03065-3283; 2010-019417-13 (EudraCT Number)
Record Dates: First submitted 2010-08-25; First posted 2010-08-30 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2016-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine; Fluticasone; MP29-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azelastine, Fluticasone (Experimental): TEST = MP29-02 = Combination product Azelastine Hydrochloride and Fluticasone Propionate nasal spray
  Interventions: Drug: Azelastine, Fluticasone
- Azelastine mono (Active Comparator): REF = AZE mono Azelastine Hydrochloride nasal spray (= essentially combination product formulation without any FLU; US AZE mono formulation as used in pivotal studies)
  Interventions: Drug: Azelastine mono
- Azelastine (Active Comparator): COMP = Astelin® Nasal Spray = AZE mono Azelastine Hydrochloride nasal spray (= US marketed product)
  Interventions: Drug: Azelastine

INTERVENTIONS:
Drug: Azelastine, Fluticasone — TEST = MP29-02 = Combination product Azelastine Hydrochloride and Fluticasone Propionate nasal spray
  Other Names: MP29-02
  Arms: Azelastine, Fluticasone
Drug: Azelastine mono — REF = AZE mono Azelastine Hydrochloride nasal spray (= essentially combination product formulation without any FLU; US AZE mono formulation as used in pivotal studies)
  Other Names: Azelastine
  Arms: Azelastine mono
Drug: Azelastine — COMP = Astelin® Nasal Spray = AZE mono Azelastine Hydrochloride nasal spray (= US marketed product)
  Other Names: Astelin®
  Arms: Azelastine

SUMMARY:
The primary objective is to assess the effect of fluticasone propionate (FLU) on the relative bioavailability (AUC0-∞) of azelastine hydrochloride (AZE) when administered as fixed AZE-FLU combination product (TEST) compared to a similar formulation without containing FLU (i.e. AZE alone; REF).

The secondary objectives are to compare the relative bioavailability (AUC0-∞) of AZE when administered either as fixed AZE-FLU combination product (TEST) or as marketed AZE product Astelin® Nasal Spray (COMP); To compare the effects of FLU on other pharmacokinetic parameters of AZE (AUC0-tlast, CL/f, Cmax, tmax, t½); To assess adverse events.

DETAILED DESCRIPTION:
This study will enrol healthy subjects. It is considered that study results are more discriminative in healthy subjects than in rhinitis patients as there are no interferences by varying rhinitis symptoms and respective differences in the status of the nasal mucosa regarding the 3 study periods.

The time schedule for plasma sampling (pre-dose and 15, 30 min, 1, 1½, 2, 2½, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 h p.a.; time refer to the end of the second spray into the second nostril of each administration) is derived from previous bioavailability study on the marketed product Astelin® Nasal Spray assuming a mean tmax of 2 to 3 h p.a. and a mean t1/2 of 22 h [L7]. Sampling times are expected to cover an AUC0-tlast above 80% of the total AUC of azelastine hydrochloride (bioanalytical detection method with a LLOQ of 2 pg/mL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects of any Ethnic origin, age from 18 to 45 years.
2. Body mass index (BMI) from 18.5 to 30.0 kg/m2.
3. Use of adequate double contraception by female with childbearing potential (i.e. women of child bearing potential using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs) or surgically sterile (documented complete hysterectomy or bi-tubal ligations; partial hysterectomy is not sufficient or vasectomised partner). It must be ensured that the male partner uses a condom during intercourse (if not surgically sterilized).
4. Use of adequate double contraception by male, who is a sexually active man and has not been surgically sterilized, must consent that he uses a condom during intercourse and ensures that his female partner practices adequate contraception (a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs) or surgically sterile (documented complete hysterectomy or bi-tubal ligations; partial hysterectomy is not sufficient).
5. Written informed consent.
6. Able to demonstrate correct nasal spray application technique at screening.

Exclusion Criteria:

1. History of allergic reaction or sensitivity to azelastine hydrochloride, fluticasone propionate or one of the excipients (e.g. benzalkoniumchloride, phenyl-ethyl alcohol).
2. Any evidence of clinically relevant acute or chronic cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, mental, neurological, or other disease at screening.
3. Positive ß-HCG pregnancy test, or established pregnancy, breast-feeding or planned pregnancy during the study.

   Lack of suitability for the study:
4. History of haemophilia or coagulation disease.
5. Significant history of orthostatic hypotension, fainting or blackouts.
6. Existence of any surgical or medical condition, which might significantly alter the absorption, distribution, metabolism, or excretion of study drug.
7. Chronic or clinically relevant acute infections (e.g. of the respiratory tract including sinusitis and rhinitis), acute rhinorrhoea or febrile disease the week before randomisation.
8. Clinical chemical, haematological or any other laboratory parameters clinically relevant outside the reference range (e.g. elevated liver enzymes, renal laboratory parameters, and coagulation abnormalities such as abnormalities of platelet count, prothrombin time, or activated partial thromboplastin time).
9. Positive results in HIV, HCV and HBsAg tests.
10. ECG abnormalities of clinical relevance, in particular abnormal prolongations of QT/QTc- or PQ-interval (i.e. QTc according to Fridericia ≥ 450 ms, PQ ≥ 220 ms).
11. Resting heart rate in the awake subject below 45 BPM or above 90 BPM, systolic blood pressure below 100 mmHg or above 145 mmHg, diastolic blood pressure above 95 mmHg.
12. Regular therapy with corticosteroids (e.g. fluticasone propionate) or antihistamines (e.g. azelastine hydrochloride).
13. Any concurrent medication or any medication within 2 weeks preceding the start of the study (single intake/use of drugs may be accepted, if judged by the investigator to have no clinical relevance and no influence on study outcome).
14. Exposure to any cytochrome P450 3A4 inhibiting or inducing drug (e.g. ritonavir, ketoconazole, itraconazole, erythromycin, rifampicin, St. John's wort (Hypericum perforatum) etc.) diets (charcoal grilled meat, brussels sprouts, broccoli) or beverages (e.g. grapefruit juice) within 14 days prior to study enrolment, or anticipated consumption of such products during that period or at any time throughout the study.
15. History of any nasal surgery or known clinically relevant abnormalities, such as rhinitis medicamentosa, polyposis, septum deviation with clinical symptoms, or nasal structural abnormalities.
16. Known perennial airway allergies. Known seasonal airway allergies which are clinically relevant acute within the last six weeks prior to the start of the study or might become acute during the study period.
17. History of malignancy within the past five years.
18. Blood donation within the last 2 months prior to the start of the study.
19. Present or history of drug or alcohol abuse within the last three years. Regular daily consumption of more than half a litre of usual beer or 0.25 L of wine per day or the equivalent quantity of approximately 30 g of alcohol in another form.
20. Current smoker or smoking during the last year.
21. Exposure to an investigational medicinal product within the last 3 months.
22. Subject reports a regular xanthine consumption of > 5 cups of coffee or black tea per day (or equivalent xanthine consumption of ≥ 500 mg xanthine per day using other products).
23. Subject is vegetarian or reports other strict dietary habits which would preclude the subject's acceptance of standardized meals
24. Lack of ability or willingness to give informed consent.
25. Lack of willingness to have personal study related data collected, archived or transmitted according to protocol.
26. Lack of willingness or inability to co-operate adequately.
27. Anticipated non-availability for study visits/procedures.
28. Vulnerable subjects (such as persons kept in detention).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effect of fluticasone propionate on the relative bioavailability of azelastine | up to 120 h post application
  Effect of fluticasone propionate (FLU) on the relative bioavailability (AUC0-∞) of azelastine hydrochloride (AZE) when administered as fixed AZE-FLU combination product (TEST) compared to a similar formulation without containing FLU (i.e. AZE alone; REF).

SECONDARY OUTCOMES:
Relative bioavailability | up to 120 h post application
  Relative bioavailability (AUC0-∞) of AZE when administered either as fixed AZE-FLU combination product (TEST) or as marketed AZE product Astelin® Nasal Spray (COMP);
Effects of fluticasone on other pharmacokinetic parameters | up to 120 h post application
  Effects of FLU on other pharmacokinetic parameters of AZE (AUC0-tlast, CL/f, Cmax, tmax, t½);
Adverse events | At and between treatment periods
  Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kolb, Study Director — MEDA Pharma GmbH & Co. KG
Locations (1):
- ClinPharmCologne, Cologne, North Rhine-Westphalia, Germany